CLINICAL TRIAL: NCT05476237
Title: Pilot Implementation of Depression Screening and Treatment for Adolescents in Mozambican Primary Care
Brief Title: Adolescent Depression Screening and Treatment in Mozambican Primary Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kathryn L. Lovero, PhD, Assistant Professor of Sociomedical Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAU3060; K01MH120258 (NIH)
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Depression; Adolescent Behavior
Keywords: adolescent depression
MeSH Terms: conditions — Depression; Adolescent Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU (Active Comparator): Psychologists or PsyTechs in mental health services of primary care clinics will provide individual psychotherapy to depressed adolescents in the TAU arm. Local mental health professionals providing depression treatment in the TAU arm will not have been trained on IPT for adults or adolescents. Also, the two Ministry of Health psychologists trained as trainers of IPT-AG will not provide treatment in the TAU Arm.
  Interventions: Behavioral: Treatment as Usual (TAU)
- IPT-AG (Experimental): Group IPT-AG will be facilitated by the trained providers at each YFHS using the IPT-AG manual adapted to the Mozambican context. Adolescents will participate in 12 weekly sessions. The first and last sessions will be one-on-one with the provider. The first session is used for the participant and provider to develop a treatment plan and the last session is to prepare for treatment termination. All other sessions will be conducted in groups of 6-8 adolescents.
  Interventions: Behavioral: Group Interpersonal Therapy for Adolescents (IPT-AG)

INTERVENTIONS:
Behavioral: Group Interpersonal Therapy for Adolescents (IPT-AG) — IPT-AG is a ten session, group therapy for adolescents. Each group contains 6-8 adolescents who attend weekly sessions together. The goals of IPT-AG are: 1) to reduce depression symptoms, and 2) to improve interpersonal relationships. Another aim of the group format is to increase adolescents' experience with positive social interactions and to reduce social isolation.
  Arms: IPT-AG
Behavioral: Treatment as Usual (TAU) — Adolescents will be administered unstructured psychotherapy in individual sessions with a trained mental health specialist (i.e., psychologist or psychiatric technician).
  Other Names: TAU
  Arms: TAU

SUMMARY:
This is a cluster-randomized pilot trial of depression screening and treatment implementation at four Youth-friendly Health Services (YFHS) in primary care clinics, two in Maputo City and two in Maputo Province. YFHS will be stratified by urbanicity, such that one YFHS in Maputo City and one YFHS in Maputo Province will be randomized to interpersonal psychotherapy (IPT)-A and the other YFHS in each location with be randomized to treatment as usual (TAU).

DETAILED DESCRIPTION:
Mental disorders are the leading cause of disability among adolescents worldwide, but only a very small minority, mostly in high-resource settings, have access to mental health care. The investigators' work is focused on understanding how to increase access to mental health care for adolescents in low-resource settings. In Mozambique, where this work is based, there are just 15 psychiatrists and 180 psychologists to serve its population of 29 million. In collaboration with local stakeholders, including governmental policymakers and primary care providers, the investigators developed a plan to implement care for adolescent depression in primary care settings. The investigators now aim to examine changes in adolescent depression and acceptability of primary care-based mental health services compared to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

1. Providers:

   1. IPT-AG Arm: YFHS staff will be included in the study if they (a) conduct screening for depression and/or group IPT-AG and (b) provide consent to participate in the study.
   2. TAU Arm: YFHS staff will be included in the study if they (a) provide referrals for adolescents suspected of having mental illness or seeking mental health services and (b) provide consent to participate in the study. Treatment providers (Psychiatric Technicians and psychologists) will be included in the study if they (a) treat adolescents referred from participating YFHS for depression and (b) provide consent to participate in the study.
2. Patients: In both study arms, adolescents attending one of the four study YFHS will be included in the study if they:

   1. are between the ages of 12-19 years;
   2. screen positive for depression;
   3. provide informed consent (ages 16 -19) or if their guardian provides informed consent and they provide assent (if ages 12-15).
3. Study centers: must be clinics that have YFHS.

Exclusion Criteria:

In both study arms, adolescents will be excluded if they:

1. are unable to participate in treatment due to acute illness; and/or
2. are unable to communicate sufficiently in Portuguese to answer inclusion questions.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
PHQ-A results | 6 months
  The Patient Health Questionnaire (PHQ)-A is a 9-item severity measure of depression for adolescents adapted from the PHQ-9. Questions ask how often an adolescent has been bothered by different depression symptoms in the past week, and responses of "not at all," "several days," "more than half the days," and "nearly every day" are given scores of 0 to 3. A total score is calculated by summing the value of all items and ranges from 0 (better outcome) to 27 (worse outcome).
IPT-AG Fidelity | 6 months
  The Group IPT-AG Fidelity Checklist is a 14-item scale that measures provider fidelity to group interpersonal therapy for adolescents. Providers are scored for superior (1), satisfactory (2), or needs improvement (3) adherence to each item on the checklist, which each represent and essential element of treatment (e.g., gives hope that depression is treatable, links depression to interpersonal problems). The score of the 14-items is averaged to compute the IPT-AG Fidelity rating (1=superior, 2=satisfactory, 3=needs improvement), with 1 indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Lovero, PhD, Principal Investigator — Columbia University
Locations (4):
- Mozambique (4):
  - Centro de Saude Alto Mae, Maputo
  - Centro de Saude Chamaculo, Maputo
  - Centro de Saude Magoanine Tendas, Maputo
  - Centro de Saude Primeiro de Maio, Maputo

IPD SHARING:
Plan to Share IPD: No